CLINICAL TRIAL: NCT05946902
Title: Comparisons of the Impact of Monotherapy With Mirabegron or Tolterodine Versus Combined Treatment With Mirabegron and Tolterodine on Autonomic Function and Bladder Blow Flow in Women With Overactive Bladder Syndrome: a Randomized Controlled Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief and Professor, Department of Obstetrics and Gynecology, Far Eastern Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 112019-F
Record Dates: First submitted 2023-07-07; First posted 2023-07-14 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Female Patients With Overactive Bladder Syndrome
MeSH Terms: interventions — Tolterodine Tartrate; mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mirabegron (Active Comparator): mirabegron 25 mg
  Interventions: Drug: mirabegron
- tolterodine (Active Comparator): tolterodine 4 mg
  Interventions: Drug: tolterodine
- combined therapy (Experimental): tolterodine 4 mg & mirabegron 25 mg
  Interventions: Drug: tolterodine , mirabegron

INTERVENTIONS:
Drug: tolterodine — tolterodine 4 mg per day
  Arms: tolterodine
Drug: mirabegron — mirabegron 25 mg per day
  Arms: mirabegron
Drug: tolterodine , mirabegron — tolterodine 4 mg and mirabegron 25 mg per day
  Arms: combined therapy

SUMMARY:
To evaluate the impact of combined therapy on the heart rate variability, compared with monotherapy in women with overactive bladder syndrome. Secondary objective is to evaluate the impact of combined therapy on bladder blood perfusion.

DETAILED DESCRIPTION:
Patients and methods:

We will conduct a prospective randomized controlled study in the outpatient clinic of Department of Obstetrics and Gynecology of Far Eastern Memorial Hospital, and will recruit 150 female patients with overactive bladder syndrome. All female patients with overactive bladder syndrome enrolled in the study will be requested to fill in the urgency severity score, the overactive bladder symptom score questionnaire, and the King's health questionnaire before taking the drug and four weeks and twelve weeks after taking the drug. In addition, measurement of heart rate variability and bladder blood perfusion will be performed.

Expected results:

We will obtain the impact of monotherapy with tolterodine or mirabegron versus combined therapy on heart rate variability and bladder blood perfusion in women with overactive bladder syndrome.

ELIGIBILITY:
Inclusion Criteria:

* >20 years old .
* female patients with overactive bladder syndrome

Exclusion Criteria:

* Cases of hypersensitivity to mirabegron or tolterodine.
* Betanley is contraindicated in the following patients: uncontrolled severe hypertension.
* Dexotol is contraindicated in the following patients: known urethral diverticulum, known bladder malignancy, patients with urinary retention and gastric retention, patients with uncontrolled narrow-angle glaucoma, patients with renal dialysis, severe renal dysfunction (ie Inulin clearance rate (GFR<30 ml/min) or liver dysfunction (i.e. liver cirrhosis), use strong CYP3A4 inhibitors such as ketoconazole.
* Patients with myasthenia gravis.
* The patient is taking drugs that interact with tolterodine or mirabegron.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Improvement of overactive bladder symptoms | 12 weeks
  Change of overactive bladder symptom score between groups

SECONDARY OUTCOMES:
Change of heart rate variability | 12 weeks
  Change of heart rate variability between groups
Change of bladder blood perfusion | 12 weeks
  Change of bladder blood perfusion between groups

OTHER OUTCOMES:
Change of quality of life | 12 weeks
  Change of King's Health Questionnaire score between groups

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No